CLINICAL TRIAL: NCT00328770
Title: De Novo Sirolimus-based Immunosuppression After Liver Transplantation for Hepatocellular Carcinoma: Long-Term Outcomes and Side Effects
Brief Title: De Novo Sirolimus-based Immunosuppression After Liver Transplantation for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Norman Kneteman, Co-zone Clinical Section Chief, Transplants/NARP, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #4279
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Liver Carcinoma
Keywords: liver transplant; hepatocellular carcinoma; sirolimus
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus based immunosuppression (Experimental): Sirolimus given intravenously or orally to achieve serum level of 12-20ug/l
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus given intravenously or orally to achieve target levels of 12-20ug/l
  Other Names: Rapamune

SUMMARY:
This study investigates whether sirolimus could decrease the rate of hepatoma recurrence after liver transplantation in high risk hepatoma patients.

DETAILED DESCRIPTION:
A total of 70 patients with HCC (mean age: 54.6 years, female/male: 12/58) received a liver transplant and were included in the study. Immunosuppression included de novo sirolimus, low-dose calcineurin inhibitor for 6 to 12 months, with short-course (3 months) or no steroids.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hepatocellular (HCC) carcinoma receiving liver transplant

Exclusion criteria:

* Patients less than 18 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 1996-12; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman M Kneteman, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Treiber G. mTOR inhibitors for hepatocellular cancer: a forward-moving target. Expert Rev Anticancer Ther. 2009 Feb;9(2):247-61. doi: 10.1586/14737140.9.2.247. PMID 19192962

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All adults receiving a liver transplant between December 1996 and March 2006 who had hepatocellular carcinoma and were treated with sirolimus as part of their immunosuppression after their transplant were included in this trial.
Groups:
- All Study Patients: All patients with hepatocellular carcinoma receiving sirolimus-based immunosuppression after liver transplantation
Period: Overall Study
Arm/Group | All Study Patients
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Patients
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 54.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 58
Region of Enrollment [Number; unit: participants]
  Canada | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Surviving at One and Four Years After Liver Transplant
Description: Percent of Patients Surviving at One & Four years after Liver Transplant was calculated
Time Frame: 1 & 4 years
Population: Percentage of patients surviving to 1 and 4 years after liver transplant was calculated for all patients
Measure: Number; unit: percentage of participants
Groups:
- Patient Survival: 1 and 4 year patient survival
Arm/Group | Patient Survival
Number analyzed (Participants) | 70
percentage of participants
  1 year patient survival | 85
  4 year patient survival | 77

2. Primary Outcome: Percentage of Participants Surviving With no Evidence of Recurrent Tumor at One and Four Years After Liver Transplant
Description: Percentage of Participants Surviving with no Evidence of Recurrent Hepatocellular Carcinoma at One and Four Years After Liver Transplant
Time Frame: 1 and 4 years
Measure: Number; unit: percentage of participants
Arm/Group | All Study Patients
Number analyzed (Participants) | 70
percentage of participants
  1 year tumor-free survival | 84
  4 year tumor-free survival | 74

3. Secondary Outcome: Sirolimus Toxicity/Intolerance
Description: Sirolimus toxicity/intolerance requiring discontinuation of sirolimus
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | All Study Patients
Number analyzed (Participants) | 70
participants | 13

ADVERSE EVENTS:
Description: Only Adverse Events related to toxicity were collected/reported.
Arm/Group | All Study Patients
Serious Adverse Events (participants affected / at risk) | 7/70
Other Adverse Events (participants affected / at risk) | 6/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Patients (N=70)
Hematological toxicity (Blood and lymphatic system disorders) | 4 (4) — Anemia defined as hemoglobin under 8 g/dL for at least one week or requiring treatment. Leucopenia defined as leukocyte counts under 3 x 10-9/L for at least 5 days or requiring granulocyte colony-stimulating factor therapy.
Delayed wound healing (Skin and subcutaneous tissue disorders) | 3 (3) — Delayed wound healing defined as a wound still requiring nursing therapy one month after surgery.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Patients (N=70)
Mouth ulcers (Gastrointestinal disorders) | 2 (2) — Oral ulcers necessitating patients being discontinued from sirolimus therapy
Dyslipidemia (Metabolism and nutrition disorders) | 1 (1) — Dyslipidemia necessitating patient have sirolimus discontinued.
Other unspecified reasons for discontinuation of sirolimus (General disorders) | 3 (3) — Reasons patients were discontinued from sirolimus therapy were not specified by the physicians who took the patients off the medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No